CLINICAL TRIAL: NCT04167475
Title: A Randomised, Double-blinded, Placebo-controlled, Parallel-group, Pilot Study to Assess the Effectiveness of the B. Longum 1714™ Strain on Subjective and Objective Sleep Quality in Healthy Men and Women
Brief Title: Effect of B. Longum 1714™ on Sleep Quality
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PrecisionBiotics Group Ltd. (Industry)
Collaborators: Nottingham Trent University (Other); Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-108
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Subjective Sleep Quality; Objective Sleep Quality
Keywords: Bifidobacterium longum 1714™; probiotic; sleep quality; PSQI; actigraphy; sleep latency; sleep efficiency
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic capsule (Experimental): The participants consume one probiotic capsule a day for 8 weeks
  Interventions: Dietary Supplement: Probiotic capsule
- Placebo capsule (Placebo Comparator): The participants consume one placebo capsule a day for 8 weeks
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Probiotic capsule — Each probiotic capsule contains 1 x 10^9 CFU B. longum 1714™ with corn starch and magnesium stearate. The probiotic capsules will be supplied by PrecisionBiotics Ltd.
  Arms: Probiotic capsule
Dietary Supplement: Placebo capsule — Each placebo capsule contains corn starch and magnesium stearate. The placebo capsules will be supplied by PrecisionBiotics Ltd.
  Arms: Placebo capsule

SUMMARY:
The aim of this study is to evaluate the effect of supplementation with the B. longum 1714™ strain on subjective and objective sleep quality in healthy participants.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group study, designed to assess the effectiveness & safety of the B. longum 1714™ strain, when consumed once daily, on sleep quality. The 8-week intervention study will be conducted in otherwise healthy participants with a Pittsburgh Sleep Quality Index (PSQI) score of greater than, or equal to 5, a HADS-A and HAD-D score less than or equal to 14 and an Insomnia Severity Index of less than 11. Participants (N=90) will be pre-screened online, then visit the study site 4 times during the course of the 8 - 10 weeks' study (2 weeks screening period, followed by 8-week intervention). The first visit will be for screening, second visit will be baseline (and start of intervention - either active or placebo), third visit will be mid-intervention, and fourth visit will be at the end of intervention. Questionnaires will be administered at visit 2, 3 and 4, and research blood and saliva will also be collected at these time points. Hair sample will be taken at visit 2 and 4 while stool sample will be collected at visit 4. Participants will wear an actigraph and fill in a sleep eDiary for the whole intervention period (from visit 2 to visit 4).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Age: 18 to 45 years of age
3. BMI < 29.9 kg/m2
4. Be willing to refrain from taking any dietary supplements or other fermented foods that contain live bacteria during the study
5. Be willing to refrain from taking any medications or preparations to improve sleep (herbal, dietary supplements, homeopathic preparations, etc.) during the study
6. If using products that contain nicotine or caffeine, agrees to continue current usage levels throughout the length of the study
7. Agrees not to undertake air travel exceeding two time zones during the period of the study
8. PSQI score of 5 and above
9. HADS-A and HADS-D score of 14 and below
10. ISI score below 11
11. Be willing to maintain stable dietary habits and physical activity levels throughout the study period
12. Be able to communicate well with the Investigator, to understand and comply with the requirements of the study and be judged suitable for the study in the opinion of the Investigator

Exclusion Criteria:

1. Less than 18 or older than 45 years of age at the time of consent
2. Use of dietary supplements or other fermented foods that contain live bacteria
3. Participant who has been on antibiotics during the past 3 months
4. Participant with a malignant disease or any concomitant end-state organ disease and/or laboratory abnormalities considered by Investigators to be risky or that could interfere with data collection
5. Participant who has a significant acute or chronic coexisting illness [cardiovascular, history of co-existing gastrointestinal, and/or gynaecological, and/or urologic pathology (e.g. colon cancer, colitis, Crohn's, celiac, IBS, endometriosis, prostate cancer) or lactose intolerance
6. Participant with inflammatory disorders (e.g. chronic fatigue syndrome, psoriasis, rheumatoid arthritis or any other inflammatory arthropathies)
7. Psychiatric diagnosis other than anxiety or depression
8. Participant who is severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year)
9. Participants who are on anxiolytics, anti-depressants, antipsychotics, anticonvulsants, centrally acting corticosteroids, opioid pain relievers, hypnotics, and/or prescribed sleep medication/ herbals (e.g. valerian)
10. Combined SF36 score of greater than +2 SD from the mean
11. Participants with a history of drug and /or alcohol abuse at the time of enrolment
12. Pregnant or lactating female, or pregnancy planned during study period
13. Participants who have undertaken air travel involving transit across two or more time zones in the month previous to the study
14. Participants who are shift workers
15. Participants with sleep disorders diagnosed by a physician such as sleep apnoea;
16. Known allergy to any of the components of the test product
17. History of illicit drug use
18. Participation in a clinical study with an investigational product within 60 days before screening, or plans to participate in another study during the study period
19. Participant has a history of non-compliance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Change in subjective sleep quality, assessed by Pittsburgh Sleep Quality Index global score | Change from baseline, assessed at 4 and 8 weeks of supplement intake
  Minimum score is 0, maximum score is 21. Higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
Change in objective sleep quality, specifically sleep latency | Change from baseline, assessed at 4 and 8 weeks of supplement intake
  Assessed by actigraph
Change in objective sleep quality, specifically sleep efficiency | Change from baseline, assessed at 4 and 8 weeks of supplement intake
  Assessed by actigraph
Change in objective sleep quality, specifically wake episodes | Change from baseline, assessed at 4 and 8 weeks of supplement intake
  Assessed by actigraph
Change in objective sleep quality, specifically wake time after sleep onset (WASO) | Change from baseline, assessed at 4 and 8 weeks of supplement intake
  Assessed by actigraph
Change in subjectively reported sleep quality, sleep latency, and sleep efficiency | Change from baseline, assessed at 4 and 8 weeks of supplement intake
  Assessed by Pittsburgh Sleep Quality Index (PSQI) subscales. Each component has a minimum score of 0, maximum score of 3. Higher scores mean worse outcome.
Change in daily sleep diaries | Change from baseline, assessed daily during 8 weeks of supplement intake
  Assess waking refreshed, night time waking and sleep quality
Change in daytime sleepiness, assessed by Epworth Sleepiness Scale | Change from baseline, assessed at 4 and 8 weeks of supplement intake
  Minimum score is 0, maximum score is 24. Higher scores indicate higher daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Murphy, PhD, Study Director — PrecisionBiotics Group Ltd.
Locations (1):
- Atlantia Food Clinical Trials Ltd., Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patterson E, Tan HTT, Groeger D, Andrews M, Buckley M, Murphy EF, Groeger JA. Bifidobacterium longum 1714 improves sleep quality and aspects of well-being in healthy adults: a randomized, double-blind, placebo-controlled clinical trial. Sci Rep. 2024 Feb 14;14(1):3725. doi: 10.1038/s41598-024-53810-w. PMID 38355674